CLINICAL TRIAL: NCT01600378
Title: Prospective Data Collection of Clinical, Pulmonary Function, Radiological, Bronchoscopic and Fibered Confocal Fluorescence Microscopy Imaging, and Pathological Characteristics in Patients With Diffuse Parenchymal Lung Diseases
Brief Title: Prospective Data Collection of Patients With Diffuse Parenchymal Lung Diseases
Status: Recruiting | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/245/Cilddatabase
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Diffuse Parenchymal Lung Diseases
Keywords: diffuse parenchymal lung disease; interstitial lung disease; idiopathic pulmonary fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to generate a prospective database of all patients evaluated for diffuse parenchymal lung diseases to provide much needed data on the various disease aetiologies, incidence and prevalence rates, clinical and radiological presentations, pathologic correlations, disease progression and response to treatment, and final outcomes in this group of patients in Singapore.

ELIGIBILITY:
Inclusion Criteria:

* All patients 21 years old and older diagnosed with suspected diffuse parenchymal lung disease (multi-lobar pulmonary infiltrates)

Exclusion Criteria:

* None

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients evaluated for diffuse parenchymal lung diseases
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-05; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Final diagnoses of patients presenting with diffuse parenchymal lung disease after complete evaluation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Su Ying Low, BMBCh, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] American Thoracic Society; European Respiratory Society. American Thoracic Society/European Respiratory Society International Multidisciplinary Consensus Classification of the Idiopathic Interstitial Pneumonias. This joint statement of the American Thoracic Society (ATS), and the European Respiratory Society (ERS) was adopted by the ATS board of directors, June 2001 and by the ERS Executive Committee, June 2001. Am J Respir Crit Care Med. 2002 Jan 15;165(2):277-304. doi: 10.1164/ajrccm.165.2.ats01. No abstract available. PMID 11790668
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066